CLINICAL TRIAL: NCT04913909
Title: Effects of Probiotic Streptococcus Salivarius Strain M18 on Oral Microbiota and Glycemic Control in Patients With Type 2 Diabetes Mellitus; A Randomized Clinical Trial
Brief Title: Effects of a Probiotic on Oral Microbiota and Glycemic Control in Type 2 Diabetics; A Randomized Clinical Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Murat Tokgoz,DDS,DrPH, Researcher, Istanbul University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: Project No. TDK-2016-20104
Record Dates: First submitted 2021-05-22; First posted 2021-06-04 (Actual); Last update posted 2021-06-04 (Actual); Status verified 2021-05

CONDITIONS: Diabetes Mellitus,Type 2; Periodontitis
Keywords: Probiotics; Diabetes mellitus; Oral microbiota; Periodontitis; Streptococcus salivarius M18
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Periodontitis; Diabetes Mellitus | interventions — Glycemic Index

STUDY DESIGN:
Intervention Model Description: The trial was a prospective randomized, double-blind, placebo-controlled intervention study.
  All patients took an oral hygiene education and were invited to give paraffin-stimulated saliva, and blood samples in the Diabetic Center. All patients were examined clinically and the results of the intraoral examination were recorded. During the intervention period of 30 nights, the participants were asked to let one Dentoblis™ or placebo lozenge slowly melt in their mouth for at least one minute before going to bed and after tooth brushing. Dentoblis™, contains 4x 109 CFU/g S. salivarius M18 strain probiotic isolated from a healthy oral microbiota.
  Neither the investigators nor the subjects were aware of the contents of the lozenges except for the research nurse, who was also responsible for keeping the codes and information confidential until after the statistical calculations. At baseline and at the end of the 30 day- intervention period, all measurements were retested.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Neither the investigators nor the subjects were aware of the contents of the lozenges except for the research nurse, who was also responsible for keeping the codes and information confidential until after the statistical calculations. Statistical analysis were performed by a blind assessor.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | US Export: No

ARMS (2):
- Dentoblis™ group (Active Comparator): In Probiotic group; Dentoblis™, as a test lozenge, contains 4 billion CFU/g S. salivarius M18 strain probiotic isolated from a healthy oral microbiota, has been utilized one lozenge a day for 30 days.
  Interventions: Dietary Supplement: Effects of an oral probiotic or placebo use on oral microbiota and glycemic index in Type 2 diabetic patients
- Placebo group (Placebo Comparator): The placebo was indistinguishable in form, size, color, smell and taste from the probiotic lozenge, but contained no bacteria and utilized one lozenge a day for 30 days . Placebo and probiotic lozenges were equivalent to 810 mg each and containing same amount of xylitol. Both were provided by the manufacturer, Bluestone Pharma GmbH, Baar, Switzerland, in equal white containers boxes, separated by production code.
  Interventions: Dietary Supplement: Effects of an oral probiotic or placebo use on oral microbiota and glycemic index in Type 2 diabetic patients

INTERVENTIONS:
Dietary Supplement: Effects of an oral probiotic or placebo use on oral microbiota and glycemic index in Type 2 diabetic patients — The participants were randomized to the interventional groups, probiotic or placebo, by the diabetes nurse. During the intervention period of 30 nights, the participants were asked to let one Dentoblis™ or placebo lozenge slowly melt in their mouth for one minute before going to bed and after tooth brushing. Dentoblis™, as a test lozenge, contains 4x109 CFU/g S. salivarius M18 strain isolated from a healthy oral microbiota and has been utilized as oral probiotic inhibiting dental caries-causing pathogens.
  The placebo is indistinguishable in form, size, color, and taste from the probiotic lozenge, but contains no bacteria. Placebo and probiotic lozenges were equivalent to 810 mg each and containing same amount of xylitol. Both were provided by the manufacturer, Bluestone Pharma GmbH, Baar, Switzerland, in equal white containers boxes, separated by production code. Neither the investigators nor the subjects were aware of the contents of the lozenges except for the research nurse.

SUMMARY:
The present study evaluated clinically the effects of a probiotic on oral microbiota and glycemic control in T2 diabetic patients with periodontal disease. The study was designed as a prospective randomized, double-blind, placebo- controlled interventional study. At baseline and at the end of the 30 day- probiotic period, all clinical, microbiological, and biochemical measurements were tested. Colony counts of oral microbiota, blood fructosamine levels and CRP were the outcomes of the study.

DETAILED DESCRIPTION:
Objectives: To investigate the effects of an oral probiotic use, containing 4 billion colony forming unit (CFU/g) Streptococcus Salivarius M18 strain (Dentoblis™), on the quantities of oral microbiota in saliva and metabolic markers of T2 diabetics such as fructosamine, C-reactive protein (CRP).

Materials and Methods: The trial was designed as a prospective randomized, double-blind, placebo- controlled interventional study. Participants were selected from type 2 diabetics with periodontitis and aged 30-65 years, who presented to the Diabetic Center in Istanbul. Totally 70 patients were randomly assigned to probiotic or placebo groups. At baseline and at the end of the 30 day-probiotic period, colony counts of oral microbiota and biochemical measurements of diabetes were assessed.

ELIGIBILITY:
Inclusion Criteria:

* being diagnosed with T2 diabetes with <10% HbA1C for at least 6 months,
* 30-65 years old patients,
* high caries activity patients with Periodontal Disease Index (PDI) scores of 2, 3, 4 and 5,
* provision of written informed consent -

Exclusion Criteria:

* patients regularly using probiotics,
* patients on corticosteroid, non-steroid anti-inflammatory, antibiotic or antibacterial mouthwash therapy,
* patients with multi-organ deficiency such as liver or kidney failure,
* patients with Immunodeficiency syndrome or on immunosuppressive therapy,
* patients with heart valve prosthesis or central venous catheter,
* patients undergoing chronic or acute disease therapy such as cancer, arthritis, influenza, flu,
* legal incapability or mental incapacity to give consent.

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2015-09-10 (Actual); Primary Completion 2017-05-18 (Actual); Study Completion 2018-03-14 (Actual)

PRIMARY OUTCOMES:
Change in the Oral Microbiota colony counts at baseline and after intervention | 30 days
  Colony counts of periodontal pathogens, S.mutans and candidas were determined 30 day after the use of the Probiotic in CFU/g
Change in blood fructosamine levels in Type 2 diabetic patients an Oral probiotic use | 30 days
  Clinical marker of Type 2 diabetics such as CRP and fructosamine were determined 30 day after the use of the Probiotic

CONTACTS AND LOCATIONS:
Overall Officials: Yeliz Mercan, PhD, Principal Investigator — Kırklareli University, Turkey

IPD SHARING:
Plan to Share IPD: Yes
All information will be available to share with other researchers
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: As of January 2022
Access Criteria: No criteria

REFERENCES:
- [Background] Burton JP, Drummond BK, Chilcott CN, Tagg JR, Thomson WM, Hale JDF, Wescombe PA. Influence of the probiotic Streptococcus salivarius strain M18 on indices of dental health in children: a randomized double-blind, placebo-controlled trial. J Med Microbiol. 2013 Jun;62(Pt 6):875-884. doi: 10.1099/jmm.0.056663-0. Epub 2013 Feb 28. PMID 23449874
- [Background] Soderling E, Hirvonen A, Karjalainen S, Fontana M, Catt D, Seppa L. The effect of xylitol on the composition of the oral flora: a pilot study. Eur J Dent. 2011 Jan;5(1):24-31. PMID 21311610